CLINICAL TRIAL: NCT03027141
Title: Pilot Study: Self-Face Recognition After Face Transplantation
Brief Title: Self-Face Recognition After Face Transplantation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-01144
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Disfigurement of Face
Keywords: Face Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Transplant Time Point (Active Comparator): Participants will be imaged in the Magnetic Resonance Imaging scanner (MRI)
  Interventions: Behavioral: Face recognition task
- Post-Transplant Time Point (Experimental): Participants will be imaged in the Magnetic Resonance Imaging scanner (MRI). Patients for whom a pre-transplant fMRI was obtained will undergo functional MRI scanning at three-points post-transplant (approximately 2 and 4 months +/- 2 months post-operation and again at 1 year +/- 3 months post-transplant).
  Interventions: Behavioral: Face recognition task

INTERVENTIONS:
Behavioral: Face recognition task — Inside the MRI scanner and during the experiment, participants will be asked to make judgments about the identity they perceived in each morphed picture.

SUMMARY:
The purpose of the proposed study is to use functional magnetic resonance imaging (fMRI) to investigate how a change in facial appearance is initially represented in brain circuits and then alters over time, as the new face becomes recognized as "me".

Investigators will try to identify areas of the brain responsible for processing and storing information about self-facial recognition; Examine how these areas of the brain respond to images of "self" and "non-self" and; Investigate how the brain responds, over time, to changes in facial recognition, particularly at time points: i) prior to facial injury, ii) post-injury but prior to facial transplantation, and iii) after receiving facial transplantation.

DETAILED DESCRIPTION:
Before surgery, investigators will compare activity in the brain when participants are looking at their pre-injury and their injured face with activity when they are looking at the persons face with whom they are familiar with. This will identify whether there are differences between how the brain responds when patients view their current facial appearance and when viewing their face before facial disfigurement. Investigators will then scan the patients post-operatively when the transplant team deems the patient ready; this will depend on reduction of post-operative swelling, improved communication with the treatment team, and patient psychological status. Activity in the brain will be compared when participants are looking at pictures of the familiar other person, with pictures of their pre-injury, pre-transplant disfigured face and pictures of their post-transplant facial appearance. Participants will be scanned again, at least two months later, with the same set of stimuli. Activity in the brain will be compared when participants look at their pre-transplant disfigured face and their new face, compared with activity when they look at the familiar other. This will allow investigators to see the differences in how the brain responds to the new facial appearance over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered from severe facial disfigurement which warrant facial transplantation and have been evaluated and approved for transplantation, will be included.

Exclusion Criteria:

* Must be be able to enter and be scanned using MRI.
* Able to give full informed consent, before each scan and throughout their time in which they are participating in the study
* Able to perform the task to a high standard and also to have no underlying conditions that may alter how they process pictures of face
* Participants must have none of the following, which cannot safely be removed without risk or discomfort while they enter the MRI unit:

  * a pacemaker
  * metal implants
  * metal that cannot be removed on their body (e.g. shrapnel, piercings)
  * metal clips
  * an artificial heart valve
  * a cochlear implant
  * drug patches
  * a contraceptive coil
  * dental plates/braces with metal in
  * hearing aids
* Participants will also be excluded on the grounds of safety and comfort inside the MRI scanner if they have one of the following underlying conditions

  * epilepsy
  * diabetes
  * heart disease
  * thermoregulatory problems (problems regulating body temperature)
  * a possibility of being pregnant
  * currently breastfeeding
* Participants will also be excluded on the grounds of MRI data quality for the following reasons:

  * history of mental illness
  * claustrophobia (discomfort in confined spaces)
  * Neurological conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Average percentage of the self in the morphs that participants judge to be "like self" for the self- face before disfigurement, | 5 Years
  This will be done by means of a series of repeated-measures analyses of variance (ANOVA statistical tests) using a computer program - the Statistical Package for the Social Sciences
Average percentage of the self in the morphs that participants judge to be "like self" for the self- face before before surgery | 5 Years
  This will be done by means of a series of repeated-measures analyses of variance (ANOVA statistical tests) using a computer program - the Statistical Package for the Social Sciences
Average percentage of the self in the morphs that participants judge to be "like self" for the self- face after surgery. | 5 Years
  This will be done by means of a series of repeated-measures analyses of variance (ANOVA statistical tests) using a computer program - the Statistical Package for the Social Sciences

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rodriguez, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States